CLINICAL TRIAL: NCT04480853
Title: A 12-month, Prospective, Multi-center Post-authorization Commitment (PAC) Study Monitoring Safety in Adult Patients With Relapsing-remitting Multiple Sclerosis Newly Initiated on Gilenya (Fingolimod) in Taiwan (SPRING)
Brief Title: Safety and Efficacy Study of Fingolimod in Taiwanese Adults (≥ 20years) With Relapsing Remitting Multiple Sclerosis
Acronym: SPRING
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFTY720DTW03
Record Dates: First submitted 2020-07-17; First posted 2020-07-21 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Multiple Sclerosis
Keywords: Fingolimod; Multiple sclerosis; Relapsing-remitting multiple sclerosis; Relapsing-remitting; Post-authorization study; Adult; MS
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fingolimod (Experimental): Open label Fingolimod 0.5 mg capsule taken once daily, oral.
  Interventions: Drug: Fingolimod

INTERVENTIONS:
Drug: Fingolimod — Fingolimod 0.5 mg QD, oral
  Other Names: FTY720

SUMMARY:
The purpose of the study is to describe the safety profile of fingolimod in the Taiwanese multiple sclerosis population. This study aims to collect the safety data in patients newly initiated on fingolimod for one year.

DETAILED DESCRIPTION:
This is a 12-month, prospective, interventional, multi-center study to monitor safety in adult patients with relapsing-remitting multiple sclerosis (RRMS) in Taiwan who based on local practice are newly starting fingolimod at the time of study entry.

Thirty-four patients will be included in this study in line with the study inclusion and exclusion criteria. After entering this study, the participants will continue to be treated for MS based on local practice. The patient will be taking fingolimod 0.5mg per day. Protocol-mandated procedures and visits for safety data collection will be conducted in addition to the required examinations according to the clinical practice.

If a patient experienced an interruption of fingolimod treatment that requires a re-evaluation of FDO, the patient will be discontinued from the study. If the treatment interruption does not require a FDO when re-starting fingolimod, the patient can continue to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

-Patients with relapsing-remitting multiple sclerosis that are fingolimod treatment naive at the time of study entry and are newly starting fingolimod based on physician judgement and according to Taiwan's fingolimod package insert (version TWI-090420)

Exclusion Criteria:

* Patients with the diagnosis of neuromyelitis optica.
* Patients who are being treated with any investigational drug at the time of study entry.
* In the last 6 months experienced myocardial infarction, unstable angina, stroke, transient ischemic attack, decompensated heart failure requiring hospitalization or Class III/IV heart failure
* A history or presence of Mobitz Type II second-degree or third-degree atrioventricular block or sick sinus syndrome, unless patient has a functioning pacemaker
* A baseline QTc interval ≥ 500 msec
* Cardiac arrhythmias requiring anti-arrhythmic treatment with Class Ia or Class III anti-arrhythmic drugs
* Patient with known immune deficiency, increased risk of opportunistic infection, severe active infection or chronic active infection.
* Patients with severe active malignancies, except for basal cell epithelioma
* Patients with severe hepatic insufficiency
* Pregnant or nursing (lactating) women or women of childbearing potential unless on contraception

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-10-12 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events of Special Interest(AESI) | First Dose Observation on the first day of taking findolimod
  The adverse events of special interest (AESI) include bradycardia and Grade 2 or higher AV block during First Dose Observation.
Number of Adverse Events of Special Interest (AESI) | Baseline up to 12 months
  The adverse events of special interest (AESI) include macular edema, abnormal liver function(ALT, AST or GGT > 5x upper normal limit), and severe lymphocytopenia(lymphocyte < 200 cells/μL).

SECONDARY OUTCOMES:
Annualized relapse reate (ARR) | Baseline up to 12 months
  The ARR will be calculated as total number of relapses experienced divided by total number of days of follow-up, and the ratio multiplied by 365. For patients withdraw from the study or switch to an alternative MS therapy prior to 12 month, the total number of days in study is defined as the number of days from baseline to the last date in study.
Change from baseline of Pulse (beats/min) | Baseline up to 12 months
  Pulse (beats/min - bpm) data will be summarized as descriptive statistics for change from baseline value (both for the period 6-hours post first dose and for further visit assessments). The frequency and percentage of notable vital sign abnormalities will be summarized. Notable criteria for pulse is > 120bpm or Increase of ≥15 bpm from baseline Or < 50bpm or Decrease of ≥15 bpm from baseline
Change from baseline of blood pressure (mmHg) | Baseline up to 12 months
  Blood pressure(BP)(mmHg) data will be summarized as descriptive statistics for change from baseline value (both for the period 6-hours post first dose and for further visit assessments). The frequency and percentage of notable vital sign abnormalities will be summarized. Notable criteria for systolic BP is ≥160 mm Hg or Increase of ≥20 mm Hg from baseline Or ≤ 90 mm Hg or Decrease of ≥ 20 mm Hg from baseline. Notable criteria for diastolic BP is ≥ 100 mmHg or Increase of ≥ 15 mm Hg from baseline Or ≤ 50 mmHg or Decrease of ≥ 15 mm Hg from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- Taiwan (5):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com